CLINICAL TRIAL: NCT07222449
Title: Wearables-and Blood-based Biomarkers-incorporated Modernisation of Circadian Rhythm Disruption Management in People Living With Alzheimer's Dementia: A Stepwise Study From Digital Inclusivity, Digital Therapy, to Digital Phenotyping and Biomarker Exploration
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Collaborators: Massachusetts General Hospital (Other); King's College London (Other)
Responsible Party: Principal Investigator, Ta-wei Guu, Consultant Psychiatrist, China Medical University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 114WFD2410317
Record Dates: First submitted 2024-12-29; First posted 2025-10-29 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer's disease; wearable device; behavioural and psychological symptoms of dementia (BPSD); blood-based biomarkersnear infrared photobiomodulation; sleep; circadian rhythm; blood-based biomarkers
MeSH Terms: conditions — Alzheimer Disease | interventions — Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: Randomised, sham-controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Photobiomodulation (Experimental): Participants allocated to this arm will receive photobiomodulation for up to 8 weeks, using a wearable headband.
  Interventions: Device: Photobiomodulation
- sham (Sham Comparator): Participants allocated to this arm will not receive photobiomodulation for up to 8 weeks, using a sham wearable headband.
  Interventions: Device: Sham (No Treatment)

INTERVENTIONS:
Device: Photobiomodulation — A near-infrared photobiomodulation wearable device.
  Arms: Photobiomodulation
Device: Sham (No Treatment) — Participants allocated to this arm will receive neglectable photobiomodulation for up to 8 weeks, using a sham wearable headband.
  Arms: sham

SUMMARY:
By 2025, Taiwan will become a super-aged society, with the number of Alzheimer's disease patients continuing to rise. However, the vast majority of dementia patients experience "behavioral and psychological symptoms of dementia" (BPSD), such as circadian rhythm disruptions and sleep disorders, which are not only difficult to assess accurately but also lack safe and effective treatments. If "wearable devices" can be accepted by elderly dementia patients, they may bring groundbreaking changes to both assessment and treatment approaches.

This project builds upon previous research and outcomes funded by the National Science and Technology Council (NSTC), the Ministry of Education, and the UK Alzheimer's Research UK (ARUK). Over four years, the project will begin by exploring "digital inclusivity" to validate the feasibility of research-grade actigraphy devices for dementia patients in Taiwan and establish a prototype research platform for wearable devices for these patients. Subsequently, in collaboration with Harvard University, the project will conduct a double-blind, randomized clinical trial to evaluate the efficacy of wearable photobiomodulation (PBM) devices in improving sleep, circadian rhythm disturbances, and other BPSD, as well as assess the user experience of integrating these two devices into a "digital therapy" model for both patients and caregivers.

Finally, the project will integrate wearable device data, patient clinical symptoms, and longitudinal results from four years of tracking the latest Alzheimer's blood-based biomarkers. In collaboration with Europe's largest remote dementia care team, RADAR-AD, the project will analyze potential digital phenotypes of dementia, explore the interactions among circadian rhythm disturbances, cognitive decline rates, and biomarkers, and establish a three-dimensional assessment model for dementia patients encompassing "clinical symptoms (both cognitive and non-cognitive)," "lifestyle and functionality," and "biological markers." This innovative approach aims to provide a more comprehensive understanding and treatment of dementia.

DETAILED DESCRIPTION:
In 2025, Taiwan will become a super-aged society, with a continuous rise in the number of people living with Alzheimer's dementia. The majority of these patients will experience "behavioural and psychological symptoms of dementia (BPSD)," such as agitation and sleep disturbances. Among these symptoms, nighttime sleep disorders and circadian rhythm disruptions not only deteriorate patients' quality of life but also impose substantial caregiving and medical costs on society, significantly increasing caregiver burden.

Currently, the assessment of such symptoms relies heavily on caregiver-reported questionnaires, which are often subjective and can only offer cross-sectional information. In Taiwan, this challenge is compounded by the fact that caregivers are often elderly individuals with cognitive decline themselves, making it difficult to accurately evaluate symptoms and develop effective treatment plans. Our previous research conducted in the UK revealed that even patients with late-stage dementia can accept to wear research-grade actigraphy with good compliance. Utilizing wearable devices for symptom assessment provides a more objective and continuous evaluation, with the analysis of emerging variables potentially contributing to a better understanding of dementia progression and the mechanisms underlying patients' circadian rhythm disturbances.

On the other hand, the treatment of circadian rhythm disruptions and sleep disorders in dementia patients heavily depends on medication. Many of these drugs lack proper indications for such use, and may increase the risk of falls and mortality. Near-infrared photobiomodulation (PBM) is a novel therapy emerged in recent years. Our team recently collaborated with Harvard University under a project funded by the Taiwanese National Science and Technology Council, successfully publishing the first findings on a "wearable PBM device" designed for home use in treating depression. The study demonstrated that the device might help improve sleep problems in elderly individuals with depression. If dementia patients can simultaneously use this device along with actigraphy devices, it could not only alleviate their sleep and circadian rhythm disturbances but also provide objective, continuous multi-dimensional symptom assessments through actigraphy and its build-in sensors.

This four-year project aims to begin with exploring "digital inclusivity," first validating the feasibility of using research-grade actigraphy among people living with Alzheimer's dementia in Taiwan, and establishing a research platform incorporating wearable devices data in this population. The investigators will then continue collaborating with Harvard University to conduct a double-blind randomized clinical trial, confirming the efficacy of wearable PBM devices in improving sleep, circadian rhythm disturbances, and other BPSD among these patients. Additionally, the investigators will assess the experiences of both patients and caregivers using a combined "digital therapy" approach involving both devices.

Finally, through the integration of the data across the four years from wearable devices, clinical symptom assessments, and the latest validated blood-based biomarkers for Alzheimer's disease, the investigators will conduct a longitudinal analysis. Collaborating with the largest European remote dementia care team, RADAR-AD, the investigators will explore potential digital phenotypes for dementia and examine the interactions between circadian rhythm disturbances, cognitive decline progression, and biomarkers. The ultimate goal is to establish a novel three-dimensional management model for dementia patients encompassing "clinical symptoms (cognitive and non-cognitive)," "lifestyle and functionality," and "biological markers."

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet the diagnostic criteria for Possible Alzheimer's Disease (Possible AD) or Probable Alzheimer's Disease (Probable AD) as defined by the National Institute on Aging-Alzheimer's Association (NIA-AA)
* Have sleep disorders, assessed either by: (1) A Pittsburgh Sleep Quality Index (PSQI) total score of greater than five, or (2) A nighttime symptom severity-frequency product score of greater than four on the Neuropsychiatric Inventory as evaluated by caregivers.
* Subjects must be community-based dementia patients who attend psychiatric outpatient clinics or participate in activities at dementia care centers or day care centers.
* Prior to inclusion, informed consent must be obtained. If cognitive impairment prevents subjects from signing, consent may be obtained from their primary caregiver (who may be a legal or professional representative).

Exclusion Criteria:

1. Severe cataracts significantly impairing visual light sensitivity.
2. Physical conditions (e.g., wrist disability) that prevent the wearing of a wrist actigraph.
3. Intracranial lesions or surgeries that have permanently disrupted circadian rhythm regulation systems (e.g., suprachiasmatic nucleus or pineal gland tumors).
4. Any other conditions deemed unsuitable for participation by the clinical physician, such as:

   * Currently experiencing acute delirium.
   * Suffering from respiratory infections, including COVID-19.
5. For Phase II participants, individuals with significant skin conditions on the head or conditions that could affect the efficacy of light therapy will be excluded. These include cases with:

   * Hemangiomas.
   * Scleroderma.
   * Psoriasis.
   * Rashes.
   * Open wounds.
   * Tattoos on the head. Additionally, individuals with head implants or those who have undergone photosensitizing drug treatments within two weeks prior to trial participation will also be excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2029-07-31 (Estimated)

PRIMARY OUTCOMES:
Sleep | 8 weeks post-treatment
  As measured by Pittsburgh Sleep Quality Index (PSQI), a questionnaire providing an overall score ranging from 0 to 21, where lower scores denote a healthier sleep quality.

IPD SHARING:
Plan to Share IPD: Undecided
We will decide if the IPD can be shared before the end of the study.

REFERENCES:
- [Result] Guu TW, Cassano P, Li WJ, Tseng YH, Ho WY, Lin YT, Lin SY, Chang JP, Mischoulon D, Su KP. Wearable, self-administered transcranial photobiomodulation for major depressive disorder and sleep: A randomized, double blind, sham-controlled trial. J Affect Disord. 2025 Mar 1;372:635-642. doi: 10.1016/j.jad.2024.12.065. Epub 2024 Dec 18. PMID 39706483
- [Result] Guu TW, Brem AK, Albertyn CP, Kandangwa P, Aarsland D, Ffytche D. Wrist-worn actigraphy in agitated late-stage dementia patients: A feasibility study on digital inclusion. Alzheimers Dement. 2024 May;20(5):3211-3218. doi: 10.1002/alz.13772. Epub 2024 Mar 18. PMID 38497216